CLINICAL TRIAL: NCT06576349
Title: Applying Self-compassion to Women's Heart Health: A Single-arm Pilot and Feasibility Study of the CALM Hearts Intervention
Brief Title: A Single-arm Pilot and Feasibility Study of the CALM Hearts Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: (# E2019:029 [HS22733])
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Self-Compassion; Physical Inactivity; Cardiovascular Diseases
Keywords: Self-compassion; physical activity; heart disease; cardiovascular disease; women; women's health; self-regulation; coping; feasibility; acceptability; pilot study; single-arm
MeSH Terms: conditions — Sedentary Behavior; Cardiovascular Diseases; Motor Activity; Heart Diseases; Self-Control | interventions — Methods

STUDY DESIGN:
Intervention Model Description: single-arm, multiple-methods, pilot and feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CALM Hearts Self-Compassion Intervention for Women at Risk for Heart Disease (Experimental): The CALM Hearts intervention will be conducted individually (i.e., one facilitator meeting with one participant) over the phone or via Zoom videoconferencing once per week for three weeks.
  Session 1 (90 minutes): Participants will learn about their CVD risk factors. The facilitator will introduce self-compassion as a tool for coping with CVD risk and adopting health behaviours. Participants will set a health behaviour goal to accomplish by intervention end.
  Sessions 2 (60 minutes) and 3 (60 minutes each): Lesson, workbook activity, and discussion on applying self-compassion to health behaviours and CVD risk.
  Participants will independently complete self-compassionate writing activities in their workbooks after Sessions 1 and 2.
  Interventions: Behavioral: Compassionate And Loving Mindset towards Heart Health Risk (CALM Hearts) Intervention

INTERVENTIONS:
Behavioral: Compassionate And Loving Mindset towards Heart Health Risk (CALM Hearts) Intervention — Self-compassion and health behaviour change intervention for women at risk for cardiovascular disease
  Other Names: CALM Hearts

SUMMARY:
The primary aims of this study are to explore the feasibility, acceptability, and safety, of the Compassionate And Loving Mindset towards heart health risk (CALM Hearts) intervention. The CALM Hearts intervention is a self-compassion intervention designed to help women cope with their cardiovascular disease (CVD) risk and adopt health behaviours. Through this research, we expect to identify opportunities to increase the feasibility and acceptability of the intervention. The secondary aims of this study are to observe the directionality of mean changes in behavioural and psychological outcomes from Pre- to Post-Intervention. We predict that all behavioural and psychological outcomes will change in a favourable direction.

Participants will be asked to complete three, weekly, intervention sessions in which they will apply self-compassion to coping with their CVD risk and increasing a chosen health behaviour. The intervention will be conducted virtually and led by a trained facilitator.

Feasibility will be assessed using pre-established criteria. After completing the intervention participants will be given the option to provide qualitative data on acceptability and safety.

Participants will also complete a battery of behaviour and psychological outcome measures at pre-intervention and one-week post-intervention

DETAILED DESCRIPTION:
Participants will be recruited via phone and email and complete an online written consent form

After consenting, participants will complete baseline measures housed on SurveyMonkey (https://www.surveymonkey.com) and will receive a fillable online workbook to complete throughout the intervention. The CALM Hearts intervention will be conducted individually (i.e., one facilitator meeting with one participant) over the phone or via Zoom videoconferencing once per week for three weeks. The intervention facilitator will be a research assistant with training in self-compassion and health psychology.

At pre-intervention, participants will complete behavioural and psychological measures (baseline survey).

In Session 1 (90 minutes), the facilitator will present report cards outlining each participant's CVD risk factors as determined by their participation in a previous study. Immediately after receiving their risk information, participants will complete an online questionnaire assessing their reactions to the CVD risk report (Session 1 measures). The facilitator will then introduce self-compassion as a tool for coping with CVD risk and adopting health behaviours. Finally, the facilitator will work with participants to set a health behaviour goal for the end of the intervention that follows the SMART goals framework (i.e., Specific, Measurable, Attainable, Realistic, and Time-bound). After Session 1, participants will receive a physical copy of their CVD risk report card in the mail.

Sessions 2 (60 minutes) and 3 (60 minutes) will apply self-compassion to participants' health behaviours and CVD risk. These sessions will include a lesson on self-compassion, a workbook activity, and a discussion with the facilitator.

After Sessions 1 and 2, participants will independently complete self-compassionate writing activities in their workbooks. We will ask participants to report the percentage of workbook activities they finish each week (0 to 100%).

One week after Session 3, participants will complete the post-intervention questionnaire and will be debriefed.

Participants will be invited to provide feedback about their experiences in the intervention via an open-ended online survey or telephone interview after the intervention concludes. These responses will contribute to assessing intervention acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were identified through the Women's Advanced Risk-assessment in Manitoba (WARM) Hearts Cohort (Rose et al., 2021).
2. Female sex is an inclusion criterion of the WARM Hearts Cohort. Therefore, all participants eligible for the CALM Hearts intervention were female.
3. Aged 55 to 75 years
4. Engaged in less than 150 minutes of weekly moderate-to-vigorous physical activity (i.e., not meeting the Canadian Physical Activity guidelines).
5. Had a moderate to high Framingham CVD risk score (D'Agostino et al., 2008), consented to future research contact after participation in the WARM Hearts Cohort.
6. Scored moderate to low on the 26-item self-compassion scale (1 to 3.6 / 5; Neff, 2003)

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility Domain 1: Recruitment | Assessed from baseline to 1-week post-intervention
  Recruitment will be assessed using the following criteria:
  * Percentage of WARM Hearts participants who are eligible. Criterion = Observe and report
  * Percentage of eligible participants who agree to participate. Criterion = Observe and report
  * Average time for enrollment, baseline questionnaire and scheduling. Criterion = 2 weeks
  * Most successful recruitment strategy. Criterion = Observe and report
Feasibility Domain 2: Retention and Adherence | Assessed from baseline to 1-week post-intervention
  Retention and adherence will be assessed using the following criteria:
  * Participant retention rate. Criterion = 80-85% at post-intervention
  * Demographics of withdrawn participants. Criterion = Observe and report
  * Reasons for withdrawal. Criterion = Observe and report
  * Session attendance. Criterion = 90%-95% attendance
  * Rates of questionnaire completion. Criterion = 80% overall completion
  * Home practice compliance. Criterion = 75% compliance
Feasibility Domain 3: Fidelity | Assessed from baseline to 1-week post-intervention
  Fidelity will be assessed using the following criteria:
  * Completion of all slides in sessions. Criterion = 90%-95% slide completion
  * Completion of topics in sessions. Criterion = 90%-95% topic completion
  * Completion of sessions within the allotted time. Criterion = 90%-95% timely completion
  * Quality of intervention delivery. Criterion = >80% fidelity as scored by the senior researcher
  * Technical difficulties with intervention delivery. Criterion = Observe and report
Feasibility Domain 4: Capacity | Assessed from baseline to 1-week post-intervention
  Capacity will be assessed using the following criteria:
  - Time required to deliver all aspects of the intervention. Criterion = Observe and report
Acceptability of the CALM Hearts Intervention | Assessed at 1-week post-intervention
  Acceptability will be assessed using post-intervention interviews and open-ended surveys administered to participants. Suggestions for increasing acceptability will be noted.
Safety of the CALM Hearts Intervention | Assessed at 1-week post-intervention
  Safety will be assessed using post-intervention interviews and open-ended surveys administered to participants. The criterion for safety = 100% safe.

SECONDARY OUTCOMES:
Self-Compassion | Assessed at baseline and 1-week post-intervention
  Self-Compassion Scale (Neff, 2003): Participants responded to 26 questions about their tendency to treat themselves with self-compassion or self-criticism using a five-point Likert scale (1 = almost never to 5 = almost always). A total score of self-compassion was determined by adding the means of all six sub-scales together and dividing by six (Neff, 2003b). Scores from this scale have good test-retest reliability (r = .80-.93) with high internal consistency (α = .92; Neff, 2003b). A sample item includes: "When things are going badly for me, I see the difficulties as part of life that everyone goes through".
Health Anxiety | Assessed at baseline and 1-week post-intervention
  Health anxiety subscale of the Multidimensional Health Questionnaire (Snell & Johnson,1997): This scale consists of five items assessing participants' health anxiety on a 5-point Likert scale (1 = not at all characteristic of me to 5 = very characteristic of me). A mean score is created to capture overall health anxiety. The Multidimensional Health Questionnaire is reliable and validated (Snell & Johnson, 1997). A sample item is: "I feel anxious when I think about my health".
Illness Self-Blame | Measured during Session 1 and at 1-week post-intervention
  Illness self-blame subscale of the Multidimensional Health Questionnaire (Snell & Johnson, 1997): This reliable and validated measure (Snell & Johnson, 1997) uses five items rated on a 5-point Likert scale (1 = not at all characteristic of me to 5 = very characteristic of me) to create a mean illness self-blame score (Snell & Johnson, 1997). A sample item is: "When I become sick or ill, I am the person to blame".
State Rumination | Measured during Session 1 and at 1-week post-intervention
  State Rumination Scale (Puterman et al., 2010): Participants responded to three items with a 5-point Likert scale (1= Not at all to 5 = A lot). A mean score was calculated to capture participants' state rumination about having a heart health risk. This scale is reliable and valid (Puterman et al., 2010). A sample item is: "Did you find it hard to stop thinking about your risk for heart disease afterwards?"
Negative Affect | Measured during Session 1 and at 1-week post-intervention
  Assessment of Negative Affect (Terry et al., 2013): Participants responded to 13 items using a 5-point Likert scale (1=not at all to 5=extremely). A mean score was calculated to assess negative affect about having a heart health risk. This measure has been used in other self-compassion research (Terry et al., 2013). A sample item is: "Rate the extent to which you feel sad about your risk for heart disease".
Health Promoting Behaviours | Assessed at baseline and 1-week post-intervention
  Health Promoting Lifestyle Profile-II (Walker & Hill-Polerecky, 1996): Participants responded to 52 questions about their engagement in various health-promoting behaviours using a 4-point Likert scale (1 = Never to 4 = Routinely). A mean score was calculated for each subscale, and a grand mean was calculated to assess overall health-promoting behaviours. This scale has demonstrated high internal consistency (Walker & Hill-Polerecky, 1996). Participants were asked to respond to the frequency with which they engage in different behaviours, such as "Choose a diet low in fat, saturated fat, and cholesterol."
Physical Activity | Assessed at baseline and 1-week post-intervention
  Short-form International Physical Activity Questionnaire (Craig et al, 2003): Participants reported the number of days they engaged in each intensity of physical activity and the average duration of each session. This is a reliable and valid measure (Lee et al., 2011). We used the International Physical Activity Questionnaire to calculate participants' weekly minutes of moderate-to-vigorous physical activity. A sample item includes: "During the last 7 days, how many bouts of 10 minutes or more did you complete of vigorous physical activities like heavy lifting, digging, aerobics, or fast bicycling?".

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Kinesiology and Recreation Management, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be made available upon request by contacting the corresponding author.
  Individual Participant Data includes anonymized raw survey data in the form of Excel spreadsheets, anonymized participant quotations from qualitative interviews (Microsoft Word documents), and researcher observations of the feasibility criteria (Microsoft Word documents and Excel Spreadsheets).
Time Frame: Anonymized data will become available in April 2021. The anonymized data will be stored indefinitely for use in future systematic reviews or meta-analyses and for access during the peer-review process.
Access Criteria: Anonymized data can be made available upon request by contacting the corresponding author.
  Data will be shared to support the conduct of future systematic reviews, meta-analyses, or other research that may build upon the CALM Hearts intervention.
  The principal investigator, Dr. Shaelyn Strachan, will review and approve/decline all requests for data sharing. Data will be shared following the University of Manitoba's data-sharing policies.

REFERENCES:
- [Background] Rose AV, Boreskie KF, Hay JL, Thompson L, Arora RC, Duhamel TA. Protocol for the WARM Hearts study: examining cardiovascular disease risk in middle-aged and older women - a prospective, observational cohort study. BMJ Open. 2021 May 25;11(5):e044227. doi: 10.1136/bmjopen-2020-044227. PMID 34035097
- [Background] Ross R, Chaput JP, Giangregorio LM, Janssen I, Saunders TJ, Kho ME, Poitras VJ, Tomasone JR, El-Kotob R, McLaughlin EC, Duggan M, Carrier J, Carson V, Chastin SF, Latimer-Cheung AE, Chulak-Bozzer T, Faulkner G, Flood SM, Gazendam MK, Healy GN, Katzmarzyk PT, Kennedy W, Lane KN, Lorbergs A, Maclaren K, Marr S, Powell KE, Rhodes RE, Ross-White A, Welsh F, Willumsen J, Tremblay MS. Canadian 24-Hour Movement Guidelines for Adults aged 18-64 years and Adults aged 65 years or older: an integration of physical activity, sedentary behaviour, and sleep. Appl Physiol Nutr Metab. 2020 Oct;45(10 (Suppl. 2)):S57-S102. doi: 10.1139/apnm-2020-0467. PMID 33054332
- [Background] Neff, K. D. (2003). The Development and Validation of a Scale to Measure Self-Compassion. Self and Identity, 2(3), 223-250. https://doi.org/10.1080/15298860309027
- [Background] Snell, W. E., & Johnson, G. (1997). The Multidimensional Health Questionnaire. American Journal of Health Behavior, 21(1), 33-42.
- [Background] Puterman, E., DeLongis, A., & Pomaki, G. (2010). Protecting us from ourselves: Social support as a buffer of trait and state rumination. Journal of Social and Clinical Psychology, 29(7), 797-820. doi:10.1521/jscp.2010.29.7.797
- [Background] Terry ML, Leary MR, Mehta S, Henderson K. Self-compassionate reactions to health threats. Pers Soc Psychol Bull. 2013 Jul;39(7):911-26. doi: 10.1177/0146167213488213. PMID 23813424
- [Background] Walker, S.N., & Hill-Polerecky, D.M. (1996). Psychometric evaluation of the Health-Promoting Lifestyle Profile II. Unpublished manuscript, University of Nebraska Medical Center.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588